CLINICAL TRIAL: NCT02040051
Title: Randomized Clinical Trial to Assess the Effect of Sound Insulation and Music Therapy on the Comfort of Mechanically Ventilated Patients Admitted to Intensive Care Unit
Brief Title: Efficacy of Sound Insulation and Music Therapy on the Comfort of Mechanically Ventilated Patients Admitted to Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Marina Mateu-Capel, Nurse Bachelor, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CEIC 13/36
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Intensive Care Units
Keywords: intensive care units; mechanical ventilation; music therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP A: Sound isolation / Music therapy (Active Comparator): * PREINTERVENTION: First hour. The patient will remain under the usual conditions of intensive care unit
  * INTERVENTION: Second hour. Sound isolation
  * INTERVENTION: Third hour. Music therapy
  * POSTINTERVENTION: Fourth hour. The patient will remain under the usual conditions of intensive care unit
  Interventions: Behavioral: Sound isolation / Music therapy
- GROUP B: Music therapy / Sound isolation (Active Comparator): * PREINTERVENTION: First hour. The patient will remain under the usual conditions of intensive care unit
  * INTERVENTION: Second hour. Music therapy
  * INTERVENTION: Third hour. Sound isolation
  * POSTINTERVENTION: Fourth hour. The patient will remain under the usual conditions of intensive care unit
  Interventions: Behavioral: Sound isolation / Music therapy

INTERVENTIONS:
Behavioral: Sound isolation / Music therapy — Sound isolation: we will used headphones Noise Candelling HI-FI Polk Audio UF 8000 Control Talk for sound isolation.
  Music therapy: we will used relaxing Zen music. Light Reiki Touch (Album: Merlin's Magic; Composer: Andreas Mock. Published in 1995 by Inner Worl Music)

SUMMARY:
The purpose of this study is to assess the effect of sound insulation and music therapy on the comfort of mechanically ventilated patients admitted to intensive care unit measured by the Bispectral Index (BIS), the Ramsay sedation scale and the Behaviour Pain Scale (BPS)

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Patients over 18 years old
* Patients with a level of consciousness BIS ≥ 50

Exclusion Criteria:

* Patients with withholding treatment
* Patients with partial or complete reduction of hearing in one or both ears
* Patients with altered mental states: psychosis, schizophrenia, paranoia, neurosis, etc.
* Patients with acute disease of the central nervous system: stroke, coma, encephalopathic process, etc.
* Patients with an axillary temperature > 37.5º

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Bispectral Index (BIS) | Up to 4 hours
Ramsay sedation scale | Up to 4 hours
Behaviour Pain Scale (BPS) | Up to 4 hours

SECONDARY OUTCOMES:
Blood pressure | Up to 4 hours
Heart rate | Up to 4 hours
Respiratory frequency | Up to 4 hours
Endotracheal aspirations | Up to 4 hours
Administration of sedatives drugs | Up to 4 hours
Administration of vasodilator and vasoconstrictor drugs | Up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marina Mateu, BSc, Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa
Locations (1):
- Fundació Althaia Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona, Spain